CLINICAL TRIAL: NCT06355440
Title: Pilot Study of Financial Navigation Program for Improving Financial Toxicity Among Breast Cancer in China
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xiaoyi Yuan, Principal Investigator, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2312288-16
Record Dates: First submitted 2024-03-28; First posted 2024-04-09 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-06

CONDITIONS: Breast Neoplasm Female; Financial Toxicity; Financial Navigation
MeSH Terms: conditions — Financial Stress

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Financial Navigation (Experimental): Participants will receive financial navigation service. During their hospitalization, participants will receive face-to-face information support with material booklets. Following discharge, weekly financial navigation information will be sent via WeChat for 1 month.
  The financial navigation encompasses comprehensive information support:
  * Strategies on patient-physician costs discussion
  * Skills for inquiring and tracking treatment-related costs
  * Basic knowledge about health insurance
  * Guidance on accessing and applying for financial assistance
  * Suggestions for returning to normal life and work
  * Strategies for holding a financial-related family meeting
  Interventions: Behavioral: Financial Navigation
- Usual Care (Active Comparator): Participants will receive usual care during hospitalization and regular follow-up after discharge. Participants have the freedom to utilize any financial resources, but financial navigators do not offer comprehensive information support. When participants actively inquire about cancer treatment-related costs or financial planning strategies, financial navigators will answer their questions.
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Financial Navigation — One-on-one information support with material booklets during hospitalization. Weekly financial navigation information will be sent via WeChat after discharge for 1 month.
  The financial navigation encompasses comprehensive information support:
  * Strategies on patient-physician costs discussion
  * Skills for inquiring and tracking treatment-related costs
  * Basic knowledge about health insurance
  * Guidance on accessing and applying for financial assistance
  * Suggestions for returning to normal life and work
  * Strategies for holding a financial-related family meeting
  Arms: Financial Navigation
Other: Usual Care — Participants will receive usual oncology care during hospitalization and regular follow-up after discharge. Participants have the freedom to utilize any financial resources, but financial navigators do not offer comprehensive information support.
  Arms: Usual Care

SUMMARY:
The goal of this pilot study is to access the feasibility and impact of a financial navigation program on improving financial toxicity among patients with breast cancer in China.

The main questions it aims to answer are:

* Is the intervention feasible and acceptable among participants?
* Does the intervention enhance participants' cost-related health literacy?
* Does the intervention reduce participants' financial toxicity?

Researchers will compare the financial navigation program with usual oncology care to preliminarily evaluate its effectiveness.

Participants will receive comprehensive information support, including:

* Strategies on patient-physician costs discussion
* Skills for inquiring and tracking treatment-related costs
* Basic knowledge about health insurance
* Guidance on accessing and applying for financial assistance
* Suggestions for returning to normal life and work
* Strategies for holding a financial-related family meeting

ELIGIBILITY:
Inclusion Criteria:

* (1) Newly diagnosed with breast cancer and undergoing surgery during this admission;
* (2) Female, age 18 years or older;
* (3) Receiving or expected to receive one or more of the following therapies: chemotherapy, radiotherapy, endocrine therapy, targeted therapy, and immunotherapy;
* (4) Eastern Cooperative Oncology Group Performance Status 0-2;
* (5) Provided informed consent to participate in this study.

Exclusion Criteria:

* (1) Diagnosed with ductal carcinoma in situ (DCIS)
* (2) Presence of any serious psychiatric disorders;
* (3) Cognitive impairments;
* (4) Difficulty in reading, writing, or communicating in Chinese.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2024-02-18 (Actual); Primary Completion 2024-03-28 (Actual); Study Completion 2024-05-07 (Actual)

PRIMARY OUTCOMES:
Eligibility rate | Approximately 1 month
  The eligibility rate will be calculated as the proportion of participants who meet the eligibility criteria among the total number of participants who will be assessed for eligibility. Reasons for participants' ineligibility will be recorded.
Consent rate | Approximately 1 month
  The consent rate will be calculated as the proportion of eligible participants who consent to participate among those who will be approached and eligible for participation. Reasons for participants' refusal to participate will be recorded.
Attrition rate | Through study completion, an average of 3 month
  The attrition rate will be calculated as the percentage of participants who withdraw from or drop out of the study after enrolment. Reasons for participants' withdrawal or dropout will be recorded.
Adherence rate | Through study completion, an average of 3 month
  The adherence rate will be calculated as the proportion of participants completing the entire program. Reasons for participants' nonadherence to the intervention will be recorded.
Patient-reported satisfaction | 1 month after discharge in Financial Navigation Arm
  Participants' satisfaction will be measured with homemade 5 item questionnaire, with higher scores indicating higher satisfaction.
Qualitative assessment of the intervention | 1 month after discharge in Financial Navigation Arm
  Participants' experiences will be captured through one-on-one, semi-structured qualitative interviews.

SECONDARY OUTCOMES:
Cost-related health literacy | Baseline, 1st month since baseline
  The cost-related health literacy will be measured with homemade 10-item questionnaire, with higher scores indicating higher cost-related health literacy.
Financial toxicity | Baseline, 1st month since baseline
  Financial toxicity will be measured with the Comprehensive Score for Financial Toxicity-Functional Assessment of Chronic Illness Therapy Version 2 (COST-FACIT-V2); lower scores (range, 0-44) indicating greater financial toxicity.
Material domain of financial toxicity | 1st month since baseline
  Material domain of financial toxicity will be measured with 2 items adapted from the Medical Expenditure Panel Survey (MEPS).
Behavioral domain of financial toxicity | 1st month since baseline
  Behavioral domain of financial toxicity will be measured by employment changes and cost-related nonadherence with 6 items adapted from MEPS and previous literature.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
We do not plan to share individual participant data due to privacy concerns and confidentiality agreements with participants.

REFERENCES:
- [Derived] Yuan X, Chen L, Sun Y, Kuang Y, Ruan J, Tang L, Qiu J, Xing W. The development and preliminary evaluation of a financial navigation program among patients with breast cancer in China. Asia Pac J Oncol Nurs. 2025 Feb 17;12:100668. doi: 10.1016/j.apjon.2025.100668. eCollection 2025 Dec. PMID 40124659